CLINICAL TRIAL: NCT06717087
Title: A Randomized Controlled Study of Acupuncture to Control Weight and Improve Pregnancy Rates in Overweight/Obese Polycystic Ovary Syndrome Patients
Brief Title: Study of Acupuncture to Control Weight and Improve Pregnancy Rates in Overweight/Obese PCOS Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2023-0156
Record Dates: First submitted 2024-11-24; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Polycystic Ovary Syndrome; Metformin; Acupuncture
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture+ intensive lifestyle intervention (Experimental): 8 weeks acupuncture+ intensive lifestyle intervention
  Interventions: Other: Acupuncture+lifestyle intervention
- metformin + intensive lifestyle intervention (Active Comparator): 8 weeks metformin treatment(metformin 500 mg three times a day with meals)+ intensive lifestyle intervention
  Interventions: Other: Metformin+lifestyle intervention

INTERVENTIONS:
Other: Acupuncture+lifestyle intervention — 8 weeks Acupuncture treatment for 2-3 times/week, 30min each time and lifestyle intervention((1) Daily intake of 1200~1500kcal of energy, dietary carbohydrate function ratio of 45-55%, lipid energy supply ratio of 20-30%, protein energy ratio of 20-30% (2) At least 150 minutes of moderate-intensity physical activity (e.g., brisk walking) per week (3) Quit smoking and drinking, and adjust psychologically)
  Other Names: group 1(Pulse Acupuncture and Moxibustion Therapeutic Instrument:KWD-808I,KWD-808II,KWD-808III )
  Arms: acupuncture+ intensive lifestyle intervention
Other: Metformin+lifestyle intervention — 8 weeks Metformin 500 mg three times a day with meals and lifestyle intervention ((1) Daily intake of 1200~1500kcal of energy, dietary carbohydrate function ratio of 45-55%, lipid energy supply ratio of 20-30%, protein energy ratio of 20-30% (2) At least 150 minutes of moderate-intensity physical activity (e.g., brisk walking) per week (3) Quit smoking and drinking, and adjust psychologically)
  Other Names: group 2
  Arms: metformin + intensive lifestyle intervention

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common cause of anovulatory infertility and is characterized by ovulatory dysfunction, increased androgens, and polycystic ovaries. The goal of this randomized control study is to compare the efficacy between acupuncture and metformin both with intensive lifestyle intervention for overweight /obese PCOS patients in weight and pregnancy rates improvement.

DETAILED DESCRIPTION:
A randomized control study is designed to compare the efficacy of acupuncture and metformin with intensive lifestyle intervention for overweight /obese PCOS patients in weight and pregnancy rate improvement. 92 patients will be enrolled from Renji Hospital affiliated with Shanghai Jiao Tong University School of Medicine and will be divided into 2 groups: acupuncture+ intensive lifestyle intervention group and metformin + intensive lifestyle intervention group. Each group used a specific treatment (shown as the group name) for 8 weeks. In this study, the role of acupuncture in improving weight control and pregnancy rate in overweight/obese PCOS patients will be evaluated, the safety and efficacy of acupuncture as well as metabolic measurements. Molecular targets and models for predicting the sensitivity and prognosis of acupuncture treatment, as well as in-depth research on the molecular mechanism of acupuncture in treating PCOS, have a guiding significance and promote the modernization of traditional medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PCOS according to the 2003 Rotterdam criteria with at least two of the following three symptoms: clinical and/or biochemical signs of hyperandrogenism (hirsutism or acne), oligomerism/amenorrhea, and/or polycystic ovaries (PCOS). Biochemical hyperandrogenism is defined as total testosterone > 2.6 nmol/L or free androgen index >7. Hirsutism is defined as an FG score ≥7. Oligomenorrhea is defined as menstrual bleeding > 35 days between menstrual periods in the past year, < 8 menstrual bleeding. Amenorrhea is < 3 cycles per year. PCO is defined by transvaginal ultrasound, where one or both ovaries ≥ 12 follicles 2-9 mm and/or ovarian volume ≥ 10 mL. Other endocrine disorders such as atypical congenital adrenal hyperplasia (17-hydroxyprogesterone <3 nmol/L), androgen-secreting tumors, or suspected Cushing syndrome are excluded.
2. Age from ≥ 20 years old (legal age of marriage) to ≤ 40 years old
3. PCOS patients: BMI ≥ 25 to ≤40kg/m2.
4. Willing to sign the consent form.

Exclusion Criteria:

1. History of severe heart disease, hematologic disease;
2. Known kidney disease (creatinine clearance rate <45mL/min), liver function ALT, AST more than 3 times the normal value, autoimmune disease or cancer;
3. Any acute disease that has the potential to alter renal function or cause tissue hypoxia;
4. Type I diabetes mellitus;
5. Medication within 12 weeks (hormonal drugs, antidepressants, other anti-diabetic drugs, contraceptives, ovulation induction drugs or other drugs that affect the trial in the judgment of the investigator);
6. Allergy to metformin hydrochloride or any excipients;
7. Blood pressure > 160/100 mm Hg;
8. Pregnancy or breastfeeding in the past three months;
9. No history of acupuncture treatment within 2 months;
10. Alcohol dependence
11. Persons with disabilities with language impairment or reduced ability to understand the information provided;
12. Those who have participated in other clinical studies within three months;
13. The man clearly diagnoses infertility-related diseases and factors.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
the level of body fat distribution | up to 8 weeks
  Compared with the baseline in two groups, the level of body fat distribution to evaluate weight control outcome
Pregnancy rates after intervention | up to 1 year
  Compared with the baseline in two groups, pregnancy rate is one of the index to evaluate reproductive outcome
Body mass index | up to 8 weeks
  Compared with the baseline in two groups, the level of body mass index to evaluate weight control outcome.

SECONDARY OUTCOMES:
Standardized TCM syndrome differentiation and classification of PCOS patients | up to 8 weeks
  Through the "tongue and pulse image, meridians, and constitution identification collection analyzer" (registration certificate number: Ji Machinery Note 20202200354), the standardized TCM syndrome differentiation and classification of PCOS patients was clarified.
Glucose metabolism | up to 8 weeks
  the area under the curve (AUC insulin), fasting insulin, glucose, computational homeostatic model assessment (HOMA)-IR and HOMA-B (i.e., isis β cell function) were calculated during the insulin-to-glucose tolerance test (OGTT)
Female menstrual pattern | up to 8 weeks
  Sex hormones, anti-mullerian hormone (AMH) and 21-day progesterone measurement
Intestinal bacteria microbiota | up to 8 weeks
  Such measurement is tested through gene and microbiota testing. Those who have taken antibiotics and live bacteria within one week are excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, MD, Principal Investigator — RenJi Hospital Department of Endocrinology and Metabolism
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China